CLINICAL TRIAL: NCT04161196
Title: Reducing Post-tonsillectomy Pain by Tonsil Pillars Suturing.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 077-19-HYMC
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Post - Tonsillectomy Pain
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with post - tonsillectomy suturing tonsil pillars (Active Comparator)
  Interventions: Procedure: tonsil pillars suturing
- patients without post - tonsillectomy suturing tonsil pillars (Placebo Comparator)
  Interventions: Procedure: tonsillectomy without tonsil pillars suturing

INTERVENTIONS:
Procedure: tonsil pillars suturing — The technique of suturing the faucial pillars is used routinely as part of uvulopalatopharyngoplasty, after performing the tonsillectomy, with postsurgical haemorrhage occurring rarely.
  Arms: patients with post - tonsillectomy suturing tonsil pillars
Procedure: tonsillectomy without tonsil pillars suturing — tonsillectomy without The technique of suturing the faucial pillars is used routinely as part of uvulopalatopharyngoplasty, after performing the tonsillectomy, with postsurgical haemorrhage occurring rarely.
  Arms: patients without post - tonsillectomy suturing tonsil pillars

SUMMARY:
comparing post-tonsillectomy pain with and without suturing tonsil pillars to investigate whether suturing tonsil pillars reduces the pain of post-tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and over.
2. patients with tonsillectomy indication due to chronic Tonsillitis.

Exclusion Criteria:

1. patients with tonsillectomy indication without chronic tonsillitis ( due to other causes).
2. chronic disease, chronic neurology disease.
3. chronic psychology disease.
4. bleeding tendency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Reducing Post-tonsillectomy Pain by Tonsil Pillars Suturing. | 1 year
  two patients' group in this study , one group will have a Tonsil pillars suturing after the tonsillectomy and the second group will not have this technique after the tonsillectomy, then patience should answer a post pain tonsillectomy questionnaire , by the questionnaire and the checkups to compare how each group affected ( using SPSS program and Statistics Methods.

IPD SHARING:
Plan to Share IPD: No